CLINICAL TRIAL: NCT03562559
Title: The Impact of Leg Movement on the Skin to Adductor Canal Distance: a Potential Cause for Catheter Displacement?
Brief Title: Skin to Adductor Canal Distance in Various Positions
Acronym: Skin to AC
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Marcus Tholin, Principal Investigator, University of British Columbia
Other Study IDs: H17-02633
Record Dates: First submitted 2018-05-29; First posted 2018-06-19 (Actual); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Knee Arthritis
Keywords: Total Knee Arthroplasty; Adductor Canal Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TKA Patients
  Interventions: Other: Measurements Using Ultrasound

INTERVENTIONS:
Other: Measurements Using Ultrasound — Ultrasound measurements will be made in 5 positions. The ultrasound probe will be measuring from a fixed external location of the thigh. The 5 positions include: external rotation, neutral, manual tissue external rotation, straight leg raise at 30 degrees and hip/knee flexion at 90 degrees.

SUMMARY:
To control pain after total knee replacement surgery a catheter (tubing) is sometimes inserted into an anatomic space containing nerves that provide sensation to parts of the knee. This space is called the adductor canal.

The catheters often stop working before we remove them for unclear reasons. The investigators think this is because the catheters become dislodged from where it was meant to be. This could be due to repeated movements of the catheter tip brought on by patients contracting their leg muscles when they ambulate or perform physio.

The investigators want to confirm this by measuring the distance from a fixed spot on the patient's thigh to the adductor canal using an ultrasound machine. The leg will be measured in various positions to simulate muscle movements. A significant change in the distance could possibly contribute to catheter dislodgement and result in catheter failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over or equal to the age of 18 years old who can understand the study protocol and are able to give consent
* Patients must be undergoing a primary total knee arthroplasty with neuraxial anaesthesia

Exclusion Criteria:

* Patients with an allergy to ultrasound transducer gel or measuring tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are recruiting patients undergoing total knee replacement. Per hospital protocol, patients will receive a spinal anesthetic and adductor canal block as part of their anesthetic regimen. After surgery, previously consented patients will have their skin to adductor canal distance measured by ultrasound in 5 different positions.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wilson, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tholin M, Wilson J, Lee S, Tang R, Sawka A, Vaghadia H. Impact of leg movement on skin-adductor canal distance: a potential cause for catheter tip displacement? Can J Anaesth. 2020 Aug;67(8):936-941. doi: 10.1007/s12630-020-01693-6. Epub 2020 May 8. PMID 32385824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients older than 18 years of age undergoing elective total knee arthroplasty who were able to give informed consent
Period: Overall Study
Arm/Group | TKA Patients
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TKA Patients
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 22
Age, Continuous [Mean (Full Range); unit: years] | 67.6 [49 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 40

OUTCOME MEASURES:

1. Primary Outcome: Skin to Adductor Canal Distance Disparity
Description: The largest distance disparity as measured from the 5 different leg positions
Time Frame: Measurements will be made on the day of surgery, no other assessment or follow up needed
Measure: Mean (90% Confidence Interval); unit: centimeters
Arm/Group | TKA Patients
Number analyzed (Participants) | 40
centimeters
  Neutral vs manual displacement distance (cm) | 1.01 [0.83 to 1.20]
  Neutral vs external rotation distance (cm) | 0.28 [0.16 to 0.39]
  Neutral vs straight leg raise distance (cm) | 0.43 [0.29 to 0.57]
  Neutral vs leg flexion distance (cm) | 0.63 [0.47 to 0.79]

ADVERSE EVENTS:
Time Frame: Adverse event date was not collected since this was an observational study
Description: There was no opportunity for adverse event since the object of the study was ultrasound measurements of anatomy.
Arm/Group | TKA Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03562559/Prot_SAP_000.pdf